CLINICAL TRIAL: NCT02273180
Title: Six-Month, Randomized, Open-Label, Parallel-group Comparison of SAR342434 to Humalog® in Adult Patients With Type 1 Diabetes Mellitus Also Using Insulin Glargine, With a 6-month Safety Extension Period
Brief Title: Comparison of SAR342434 to Humalog as the Rapid Acting Insulin in Adult Patients With Type 1 Diabetes Mellitus Also Using Insulin Glargine
Acronym: SORELLA1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC12619; 2013-002945-12 (EudraCT Number); U1111-1131-5038 (Other: UTN)
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Results first posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2017-12

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — SAR342434; Insulin Lispro; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SAR342434 (Experimental): SAR342434 before meals intake on top of once daily (QD) Insulin Glargine, up to Week 52.
  Interventions: Drug: SAR342434; Drug: Insulin glargine HOE901
- Humalog (Active Comparator): Humalog before meals intake on top of QD Insulin Glargine, up to Week 52.
  Interventions: Drug: Humalog; Drug: Insulin glargine HOE901

INTERVENTIONS:
Drug: SAR342434 — SAR342434 100 U/mL (dose range of 1 Unit to 80 Units) self-administered by deep subcutaneous (SC) injection, immediately (within 5-10 minutes) before meal intake. Dose adjusted to achieve a 2-hour post prandial plasma glucose (PPG) in range of 6.7 to 8.9 mmol/L (120 to 160 mg/dL) while avoiding hypoglycemia.
  Arms: SAR342434
Drug: Humalog — Humalog 100 U/mL (dose range of 1 unit to 60 units) self-administered by deep SC injection, immediately (within 5-10 minutes) before meal intake. Dose adjusted to achieve a 2 hour PPG in range of 6.7 to 8.9 mmol/L (120 to 160 mg/dL) while avoiding hypoglycaemia.
  Other Names: Insulin Lispro
  Arms: Humalog
Drug: Insulin glargine HOE901 — Insulin glargine 100 U/mL injected QD subcutaneously consistent with the local label. Doses adjusted to achieve glycemic target for fasting, preprandial plasma glucose (SMPG) between 4.4 to 7.2 mmol/L (80 to 130 mg/dL) without hypoglycemia.
  Other Names: Lantus

SUMMARY:
Primary Objective:

To demonstrate non-inferiority of SAR342434 versus Humalog in glycated haemoglobin A1c (HbA1c) change from baseline to Week 26 in participants with type 1 diabetes mellitus (T1DM) also using insulin glargine.

Secondary Objectives:

To assess the immunogenicity of SAR342434 and Humalog in terms of positive/negative status and antibody titers at baseline and during the course of the study.

To assess the relationship of anti-insulin antibodies with efficacy and safety including during the safety extension.

To assess the efficacy of SAR342434 and Humalog in terms of proportion of participants reaching target HbA1c (<7%), Fasting plasma glucose (FPG), self-measured plasma glucose (SMPG) profiles, and insulin dose.

To assess safety of SAR342434 and Humalog.

DETAILED DESCRIPTION:
The study consisted of a:

* Up to 2 weeks screening period
* 26-week treatment period
* 26-week comparative safety extension period
* 1-day follow-up period
* The maximum study duration would be 54 weeks per participant and a 1-day safety follow-up

ELIGIBILITY:
Inclusion criteria:

* Participants with T1DM diagnosed for at least 12 months and had been treated with insulin glargine and Humalog or Novolog®/Novo Rapid® (at least 3 times daily before each meal) in the 6 months prior to the screening visit.
* Written informed consent.

Exclusion criteria:

* At screening visit, age under legal age of adulthood.
* HbA1c <7.0% or >10% at screening.
* Diabetes other than T1DM.
* Status post pancreatectomy.
* Status post pancreas and/or islet cell transplantation.
* Pregnancy and lactation.
* Women of childbearing potential not protected by highly effective contraceptive method of birth control.
* Less than 1 year on continuous insulin treatment.
* Use of insulin pump in the last 6 months before screening visit.
* Use of glucose lowering treatments other than insulin including non-insulin injectable peptides in the last 6 months prior to screening visit.
* Use of insulin other than insulin glargine and Humalog or Novolog/Novo Rapid as part of a multiple injection regimen (3 to 4 injections per day) in the last 6 months before screening visit. Liprolog® is a European Union approved insulin lispro and is allowed in those countries where it is marketed.
* Hospitalization for diabetic ketoacidosis in the last 6 months before screening visit.
* Unstable proliferative diabetic retinopathy or any other rapidly progressive diabetic retinopathy or macular edema likely to require treatment (eg, laser, surgical treatment, or injectable drugs) during the study period.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (89):
- United States (47):
  - Investigational Site Number 840049, Tucson, Arizona
  - Investigational Site Number 840016, Bell Gardens, California
  - Investigational Site Number 840048, Chula Vista, California
  - Investigational Site Number 840046, Concord, California
  - Investigational Site Number 840039, Fresno, California
  - Investigational Site Number 840028, La Jolla, California
  - Investigational Site Number 840022, Ventura, California
  - Investigational Site Number 840003, Denver, Colorado
  - Investigational Site Number 840037, Denver, Colorado
  - Investigational Site Number 840005, Bradenton, Florida
  - Investigational Site Number 840050, Miami, Florida
  - Investigational Site Number 840042, Miami, Florida
  - Investigational Site Number 840061, Miami Lakes, Florida
  - Investigational Site Number 840057, Miami Lakes, Florida
  - Investigational Site Number 840006, New Port Richey, Florida
  - Investigational Site Number 840013, North Miami Beach, Florida
  - Investigational Site Number 840031, Port Charlotte, Florida
  - Investigational Site Number 840036, Atlanta, Georgia
  - Investigational Site Number 840045, Roswell, Georgia
  - Investigational Site Number 840020, Idaho Falls, Idaho
  - Investigational Site Number 840019, Chicago, Illinois
  - Investigational Site Number 840033, Chicago, Illinois
  - Investigational Site Number 840012, McHenry, Illinois
  - Investigational Site Number 840004, Des Moines, Iowa
  - Investigational Site Number 840043, Marrero, Louisiana
  - Investigational Site Number 840021, Metairie, Louisiana
  - Investigational Site Number 840038, Baltimore, Maryland
  - Investigational Site Number 840014, Rockville, Maryland
  - Investigational Site Number 840060, Great Falls, Montana
  - Investigational Site Number 840026, Omaha, Nebraska
  - Investigational Site Number 840040, Omaha, Nebraska
  - Investigational Site Number 840015, Albuquerque, New Mexico
  - Investigational Site Number 840054, Albuquerque, New Mexico
  - Investigational Site Number 840059, Mineola, New York
  - Investigational Site Number 840030, Burlington, North Carolina
  - Investigational Site Number 840051, Greenville, North Carolina
  - Investigational Site Number 840062, Wilmington, North Carolina
  - Investigational Site Number 840018, Gallipolis, Ohio
  - Investigational Site Number 840007, Dakota Dunes, South Dakota
  - Investigational Site Number 840027, Rapid City, South Dakota
  - Investigational Site Number 840041, Dallas, Texas
  - Investigational Site Number 840029, Dallas, Texas
  - Investigational Site Number 840034, Dallas, Texas
  - Investigational Site Number 840002, Houston, Texas
  - Investigational Site Number 840011, Chesapeake, Virginia
  - Investigational Site Number 840023, Tacoma, Washington
  - Investigational Site Number 840009, Milwaukee, Wisconsin
- France (4):
  - Investigational Site Number 250002, Corbeil-Essonnes
  - Investigational Site Number 250005, Mantes-la-Jolie
  - Investigational Site Number 250003, Montpellier
  - Investigational Site Number 250001, Vandœuvre-lès-Nancy
- Germany (8):
  - Investigational Site Number 276001, Berlin
  - Investigational Site Number 276004, Dortmund
  - Investigational Site Number 276006, Hanover
  - Investigational Site Number 276002, Heidelberg
  - Investigational Site Number 276003, Neumünster
  - Investigational Site Number 276008, Pirna
  - Investigational Site Number 276007, Potsdam
  - Investigational Site Number 276005, Sulzbach-Rosenberg
- Hungary (7):
  - Investigational Site Number 348002, Budapest
  - Investigational Site Number 348005, Budapest
  - Investigational Site Number 348003, Budapest
  - Investigational Site Number 348011, Budapest
  - Investigational Site Number 348010, Budapest
  - Investigational Site Number 348001, Budapest
  - Investigational Site Number 348007, Debrecen
- Japan (6):
  - Investigational Site Number 392006, Chūōku
  - Investigational Site Number 392003, Higashiosaka-Shi
  - Investigational Site Number 392004, Izumisano
  - Investigational Site Number 392005, Kamakura-Shi
  - Investigational Site Number 392001, Shinjuku-Ku
  - Investigational Site Number 392002, Yamato-Shi
- Poland (5):
  - Investigational Site Number 616005, Krakow
  - Investigational Site Number 616001, Poznan
  - Investigational Site Number 616003, Szczecin
  - Investigational Site Number 616002, Warsaw
  - Investigational Site Number 616004, Zabrze
- Russia (7):
  - Investigational Site Number 643003, Moscow
  - Investigational Site Number 643004, Saint Petersburg
  - Investigational Site Number 643001, Saint Petersburg
  - Investigational Site Number 643005, Saint Petersburg
  - Investigational Site Number 643006, Samara
  - Investigational Site Number 643002, Saratov
  - Investigational Site Number 643007, Tomsk
- Spain (5):
  - Investigational Site Number 724002, A Coruña
  - Investigational Site Number 724001, Cáceres
  - Investigational Site Number 724004, Lleida
  - Investigational Site Number 724005, Málaga
  - Investigational Site Number 724003, Sabadell

REFERENCES:
- [Background] Garg SK, Wernicke-Panten K, Rojeski M, Pierre S, Kirchhein Y, Jedynasty K. Efficacy and Safety of Biosimilar SAR342434 Insulin Lispro in Adults with Type 1 Diabetes Also Using Insulin Glargine-SORELLA 1 Study. Diabetes Technol Ther. 2017 Sep;19(9):516-526. doi: 10.1089/dia.2017.0117. Epub 2017 Aug 30. PMID 28722480

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 89 centres in 8 countries. A total of 668 participants were screened between 28 October 2014 and 04 June 2015, of which 161 participants were screen failures. Screen failures were mainly due to glycated hemoglobin A1c (HbA1c) level <7.0% or >10% at the screening visit.
Pre-assignment Details: A total of 507 participants were randomized in the study. Randomization was stratified by HbA1c at the screening visit (<8%, >=8%), prior use of Humalog/Liprolog (Yes, No) and geographical region (Non-Japan, Japan). Assignment to arms was done centrally using interactive voice/web response system in 1:1 ratio (SAR342434: Humalog).
Groups:
- SAR342434: SAR342434 100 Units(U)/mL subcutaneous (SC) injection, before meals intake on top of once daily (QD) Insulin Glargine, up to Week 52.
- Humalog: Humalog 100 U/mL SC injection, before meals intake on top of QD Insulin Glargine, up to Week 52.
Period: Overall Study
Arm/Group | SAR342434 | Humalog
Started | 253 | 254
Treated | 252 | 254
Completed | 226 | 235
Not Completed | 27 | 19
Not completed — Adverse Event | 2 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 1 | 7
Not completed — Randomized but not treated | 1 | 0
Not completed — Hypoglycemia(not reported as serious AE) | 1 | 0
Not completed — Other than specified above | 21 | 10

BASELINE CHARACTERISTICS:
Groups:
- SAR342434: SAR342434 100 U/mL SC injection, before meals intake on top of QD Insulin Glargine, up to Week 52.
- Total: Total of all reporting groups
Arm/Group | SAR342434 | Humalog | Total
Number analyzed (Participants) | 253 | 254 | 507
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (14.5) | 42.6 (13.9) | 43.0 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 101 | 205
  Male | 149 | 153 | 302
Previous mealtime insulin type [Count of Participants; unit: Participants]
  Humalog/Liprolog | 155 | 152 | 307
  NovoLog/NovoRapid | 95 | 95 | 190
  Both Humalog/Liprolog and NovoLog/NovoRapid | 3 | 7 | 10
Randomization Strata of Screening HbA1c [Count of Participants; unit: Participants]
  <8 % | 99 | 99 | 198
  >=8% | 154 | 155 | 309
Randomization strata of geographical region [Count of Participants; unit: Participants]
  Japan | 31 | 30 | 61
  Non-Japan | 222 | 224 | 446
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.2 (4) | 25.8 (4.1) | 26.0 (4.1)
Duration of Diabetes Type 1(T1DM) [Mean (Standard Deviation); unit: years] | 19.53 (12.63) | 18.57 (11.99) | 19.05 (12.31)
Average Daily Basal Insulin Dose [Mean (Standard Deviation); unit: Units (U)/kg] — Population: Number of participants analyzed = participants with available data for specified measure.
  Units (U)/kg
    number analyzed (Participants) | 245 | 245 | 490
    (all) | 0.339 (0.195) | 0.33 (0.141) | 0.335 (0.170)
Average Daily Mealtime Insulin Dose [Mean (Standard Deviation); unit: U/kg] — Population: Number of participants analyzed = participants with available data for specified measure.
  U/kg
    number analyzed (Participants) | 241 | 244 | 485
    (all) | 0.364 (0.175) | 0.355 (0.168) | 0.360 (0.172)
Average Daily Total Insulin Dose [Mean (Standard Deviation); unit: U/kg] — Population: Number of participants analyzed = participants with available data for specified measure.
  U/kg
    number analyzed (Participants) | 239 | 241 | 480
    (all) | 0.704 (0.309) | 0.685 (0.242) | 0.695 (0.278)
Glycated Haemoglobin (HbA1c %) [Mean (Standard Deviation); unit: percentage of hemoglobin] | 8.07 (0.79) | 7.99 (0.64) | 8.03 (0.72)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 26
Description: Change in HbA1c was calculated by subtracting baseline value from Week 26 value. Adjusted least square means and standard errors were obtained from a mixed-effect model with repeated measures (MMRM) to account for missing data, using all post-baseline HbA1c data available during the main 6-month period and adequate contrasts at Week 26.
Time Frame: Baseline, Week 26
Population: Analysis was performed on intent-to-treat (ITT) population that included all randomized participants, irrespective of compliance with the study protocol and procedures. Here, number of participants analyzed = participants with at least one post-baseline HbA1c assessment during the main 6-month period.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | SAR342434 | Humalog
Number analyzed (Participants) | 247 | 249
percentage of HbA1c | -0.42 (0.051) | -0.47 (0.05)
Statistical Analysis 1: Comparison: SAR342434 vs Humalog; Analysis was performed using a MMRM approach with treatment groups, randomization strata, visits and treatment-by-visit interaction as fixed categorical effects, and baseline HbA1c value and baseline HbA1c value-by-visit interaction as continuous fixed covariates. An unstructured correlation matrix was used to model within-participant errors; Test type: Non-Inferiority — Non-inferiority of SAR342434 over Humalog was demonstrated if upper bound of 2-sided 95% confidence interval(CI) of difference between SAR342434 & Humalog was <0.3%.Inverse non-inferiority of Humalog over SAR342434 was tested using hierarchical step-down testing procedure:if non-inferiority of SAR342434 over Humalog was demonstrated,then inverse non-inferiority of Humalog over SAR342434 was tested, demonstrated if lower bound of 2-sided 95%CI of difference between SAR342434 & Humalog was >-0.3%; Least Square (LS) Mean Difference = 0.06, 95% CI 2-sided [-0.084 to 0.197], Standard Error of Mean 0.071 — SAR342434 vs. Humalog

2. Secondary Outcome: Percentage of Participants With HbA1c <7.0% at Week 26
Description: Participants who had no available assessment for HbA1c at Week 26 were considered as non-responders.
Time Frame: Week 26
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | SAR342434 | Humalog
Number analyzed (Participants) | 253 | 254
percentage of participants | 22.5 | 21.7

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 26
Description: Change in FPG was calculated by subtracting baseline value from Week 26 value. Adjusted least squares means and standard errors were obtained from a MMRM approach to account for missing data, using all post-baseline FPG data available during the main 6-month period and adequate contrasts at Week 26.
Time Frame: Baseline, Week 26
Population: Analysis was performed on ITT population. Here, number of participants analyzed = participants with at least one post-baseline FPG assessment during the main 6-month period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | SAR342434 | Humalog
Number analyzed (Participants) | 240 | 242
mmol/L | -0.46 (0.248) | -0.62 (0.248)

4. Secondary Outcome: Change in Mean 24-Hour Plasma Glucose Concentration From Baseline to Week 26
Description: Mean 24-hour plasma glucose concentration was calculated based on 7-point self-measured plasma glucose (SMPG) profiles with plasma glucose measurements before and 2-hours after each main meal and at bedtime. Mean 24-hour plasma glucose concentration was calculated for each profile and then averaged across profiles performed in week before a visit. Change in mean 24-hour plasma glucose concentration was calculated by subtracting baseline value from Week 26 value. Adjusted least squares means and standard errors were obtained from a MMRM to account for missing data, using all post-baseline data available during the main 6-month period and adequate contrasts at Week 26.
Time Frame: Baseline, Week 26
Population: Analysis was performed on ITT population. Here, number of participants analyzed = participants with at least one post-baseline mean 24-hour plasma glucose concentration assessment during the main 6-month period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | SAR342434 | Humalog
Number analyzed (Participants) | 216 | 207
mmol/L | -0.23 (0.145) | -0.49 (0.148)

5. Secondary Outcome: Change in Post Prandial Plasma Glucose (PPG) Excursion From Baseline to Week 26
Description: Plasma glucose excursions were calculated at breakfast, lunch and dinner for each 7-point SMPG profile, as 2-hour PPG minus plasma glucose value obtained 30 minutes prior to start of the meal. Values of plasma glucose excursions at each visit were then calculated as average across the profiles performed in the week before the visit. Change in PPG excursions was calculated by subtracting baseline value from Week 26 value. Adjusted least squares means and standard errors were obtained from a MMRM to account for missing data, using all post-baseline data available during the main 6-month period and adequate contrasts at Week 26.
Time Frame: Baseline, Week 26
Population: Analysis was performed on ITT population. Here, number analyzed in each row = participants with at least one post-baseline data during the main 6-month period for specified categories.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | SAR342434 | Humalog
Number analyzed (Participants) | 253 | 254
mmol/L
  At breakfast: number analyzed (Participants) | 205 | 198
  At breakfast | -0.46 (0.297) | 0.19 (0.297)
  At lunch: number analyzed (Participants) | 207 | 193
  At lunch | 0.14 (0.298) | -0.26 (0.309)
  At dinner: number analyzed (Participants) | 208 | 190
  At dinner | 0.48 (0.308) | 0.56 (0.324)

6. Secondary Outcome: Number of Hypoglycemia Events (Any Hypoglycemia, Documented Symptomatic Hypoglycemia and Severe Hypoglycemia) Per Participant-Year
Description: Number of treatment-emergent hypoglycemia events per participant-year of exposure were reported. Severe hypoglycemia was an event in which the participant required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Documented symptomatic hypoglycemia was an event during which typical symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of <=70 mg/dL (3.9 mmol/L). Hypoglycemic episodes with plasma glucose of 54 mg/dL (<3.0 mmol/L) were also analyzed.
Time Frame: First dose of study drug up to 1 day after the last dose administration (maximum treatment exposure: 400 days)
Population: Analysis was performed on safety population that included all participants randomized and exposed to at least 1 dose of investigational medicinal product (IMP) (SAR342434 or Humalog), regardless of the amount of treatment administered.
Measure: Number; unit: events per participant-year
Arm/Group | SAR342434 | Humalog
Number analyzed (Participants) | 252 | 254
events per participant-year
  Any hypoglycemia | 90.71 | 92.7
  Severe hypoglycemia | 0.73 | 0.28
  Documented Symptomatic Hypoglycemia (<=3.9 mmol/L) | 29.36 | 31.37
  Documented Symptomatic Hypoglycemia (<3.0 mmol/L) | 6.29 | 6.85

7. Secondary Outcome: Percentage of Participants With Hypersensitivity Reactions and Injection Site Reactions
Description: Percentage of participants with hypersensitivity reactions and injection site reactions were reported.
Time Frame: First dose of study drug up to 1 day after the last dose administration (maximum treatment exposure: 400 days)
Population: Analysis was performed on safety population.
Measure: Number; unit: percentage of participants
Arm/Group | SAR342434 | Humalog
Number analyzed (Participants) | 252 | 254
percentage of participants
  Any hypersensitivity reactions | 6 | 6.3
  Any injection site reactions | 1.2 | 1.2

8. Secondary Outcome: Percentage of Participants With Treatment Emergent Anti-insulin Antibodies (AIAs)
Description: Participants with treatment-emergent AIA (incidence) were reported (as participants with treatment-boosted or treatment-induced AIAs). Participants with treatment-induced AIAs were those who developed AIA following IMP administration (participants with at least one positive AIA sample at any time during on-treatment period, in those participants without pre-existing AIA or with missing baseline sample). Participants with treatment-boosted AIAs were those with pre-existing AIAs that were boosted to a significant higher titer following IMP administration (participants with at least one AIA sample with at least a 4-fold increase in titers compared to baseline value at any time during on-treatment period, in those participants with pre-existing AIA).
Time Frame: First dose of study drug up to 1 day after the last dose administration (maximum treatment exposure: 400 days)
Population: Analysis was performed on anti-insulin antibody population that included all participants randomized and exposed to at least 1 dose of IMP (SAR342434 or Humalog) with at least one AIA sample available for analysis during the 12-month on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | SAR342434 | Humalog
Number analyzed (Participants) | 248 | 252
percentage of participants | 22.6 | 24.2

9. Other Pre Specified Outcome: Change in Daily Insulin Dose From Baseline to Week 26 and Week 52
Description: Change in daily insulin dose (basal, mealtime and total) was calculated by subtracting baseline value from Week 26 and Week 52 values respectively.
Time Frame: Baseline, Week 26, Week 52
Population: Analysis was performed on safety population. Here, number analyzed in each row = participants with available data for specified categories.
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | SAR342434 | Humalog
Number analyzed (Participants) | 252 | 254
U/kg
  Basal insulin dose at Week 26: number analyzed (Participants) | 223 | 229
  Basal insulin dose at Week 26 | 0.03 (0.236) | 0.014 (0.06)
  Mealtime insulin dose at Week 26: number analyzed (Participants) | 217 | 222
  Mealtime insulin dose at Week 26 | 0.005 (0.112) | -0.005 (0.089)
  Total insulin dose at Week 26: number analyzed (Participants) | 215 | 220
  Total insulin dose at Week 26 | 0.019 (0.134) | 0.01 (0.111)
  Basal insulin dose at Week 52: number analyzed (Participants) | 199 | 209
  Basal insulin dose at Week 52 | 0.046 (0.364) | 0.013 (0.066)
  Mealtime insulin dose at Week 52: number analyzed (Participants) | 192 | 203
  Mealtime insulin dose at Week 52 | 0.018 (0.117) | 0.007 (0.104)
  Total insulin dose at Week 52: number analyzed (Participants) | 191 | 200
  Total insulin dose at Week 52 | 0.039 (0.135) | 0.019 (0.127)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (maximum treatment exposure: 400 days) regardless of seriousness or relationship to investigational product.
Description: Reported AEs and deaths are treatment emergent AEs that is AEs that developed/worsened or became serious and deaths that occurred during the 'on treatment period' (time from first injection of IMP up to 1 day after the last injection of IMP). Analysis was performed on safety population.
Arm/Group | SAR342434 | Humalog
All-Cause Mortality (participants affected / at risk) | 1/252 | 0/254
Serious Adverse Events (participants affected / at risk) | 20/252 | 19/254
Other Adverse Events (participants affected / at risk) | 46/252 | 41/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAR342434 (N=252) | Humalog (N=254)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Cardiac death (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 3 | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrong drug administered (Injury, poisoning and procedural complications) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ventricle dilatation (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 0 | 1
Hypoglycaemic seizure (Nervous system disorders) | 0 | 1
Hypoglycaemic unconsciousness (Nervous system disorders) | 6 | 6
Migraine (Nervous system disorders) | 1 | 0
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pregnancy of partner (Social circumstances) | 0 | 1
Gastrectomy (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SAR342434 (N=252) | Humalog (N=254)
Nasopharyngitis (Infections and infestations) | 33 | 28
Upper respiratory tract infection (Infections and infestations) | 15 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.